CLINICAL TRIAL: NCT07306494
Title: Compound Ciwujia Granules in the Treatment of Insomnia: a Multi-center, Double-blind, Double-dummy, Randomized Controlled Trial
Brief Title: Compound Ciwujia Granules in the Treatment of Insomnia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hui Zhu (Other)
Responsible Party: Sponsor-Investigator, Hui Zhu, Resident Physician, Hubei Hospital of Traditional Chinese Medicine
Organization: Hubei Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBZY2024-C61-03
Record Dates: First submitted 2025-11-27; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Insomnia Disorder
Keywords: Compound Ciwujia Granules; multicenter; randomized controlled trial; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Estazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment of Compound Ciwujia Granules (Experimental)
  Interventions: Drug: Compound Ciwujia Granules group
- Treatment of estazolam (Active Comparator)
  Interventions: Drug: Estazolam
- Combined treatment of Compound Ciwujia Granules and estazolam (Other)
  Interventions: Drug: Compound Ciwujia Granules and estazolam

INTERVENTIONS:
Drug: Compound Ciwujia Granules group — Compound Ciwujia Granules for 4 consecutive weeks combined with placebo of estazolam for 4 consecutive weeks
  Arms: Treatment of Compound Ciwujia Granules
Drug: Estazolam — estazolam for 2 consecutive weeks + placebo of estazolam for 2 consecutive weeks combined with placebo of Compound Ciwujia Granules for 4 consecutive weeks
  Arms: Treatment of estazolam
Drug: Compound Ciwujia Granules and estazolam — Compound Ciwujia Granules for 4 consecutive weeks combined with estazolam for 2 consecutive weeks+ placebo of estazolam for 2 consecutive weeks
  Arms: Combined treatment of Compound Ciwujia Granules and estazolam

SUMMARY:
The goal of this multicenter, double-blind, double-dummy, randomized controlled trial was to examine the efficacy and safety of Compound Ciwujia Granules in the treatment of chronic insomnia. A total of 1200 participants with chronic insomnia were randomly assigned to receive one of the three treatment for 4 consecutive weeks: Compound Ciwujia Granules + placebo of estazolam, estazolam + placebo of estazolam + placebo of Compound Ciwujia Granules, or Compound Ciwujia Granules + estazolam + placebo of estazolam. Outcomes were assessed at 2 weeks, 4 weeks, 8 weeks, and 12 weeks. The main questions it aims to answer are:

1. Are there any significant differences between groups regarding changes in Pittsburgh Sleep Quality Index (PSQI) score, Insomnia Severity Index (ISI) score, subjective sleep latency, sedative and hypnotics use, improvement in sleep maintenance, Hamilton Depression Scale (HAMD-17) score, Hamilton Anxiety Scale (HAMA-14) score, Flinders Fatigue Scale (FFS) score, and constitution classification/insomnia pattern score of traditional Chinese medicine after 4 weeks' treatment, and follow-up at 8 weeks and 12 weeks.
2. Is the Compound Ciwujia Granules a safe method for chronic insomnia treatment in adults?

DETAILED DESCRIPTION:
The investigators aimed to examine the efficacy and safety of Compound Ciwujia Granules in the treatment of chronic insomnia in a multicenter, double-blind, double-dummy, randomized controlled clinical trial. Eligible participants were adults aged 40-75 years who had insomnia disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition [DSM5]) or self-reported history of disturbed sleep, diagnosis of "deficiency of the heart and the spleen pattern" or "Qi deficiency of the heart and gallbladder pattern" according to the guidelines for Integrated Traditional Chinese and Western Medicine Treatment of Insomnia Disorders 2023, baseline Pittsburgh Sleep Quality Index (PSQI) score ≥ 8. The exclusion criteria were (1) self-reported allergy symptoms to any of the ingredients; (2) serious physical sickness; (3) a history of suicidal ideation or attempt, acute or chronic psychiatric condition not controlled by therapy; (4) baseline HAMD-17 score ≥17 or HAMA-14 score ≥14;(5) pregnant women; (6) history of drugs or alcohol abuse/dependence; (7) presence of other sleep disorders including sleep apnoea, restless legs syndrome; (8) night, morning or rotating shift work; (9) participation in concurrent clinical trials. The primary outcome was the change in Pittsburgh Sleep Quality Index (PSQI) score after 4 weeks' treatment. The secondary outcomes were changes in Insomnia Severity Index (ISI) score, subjective sleep latency, sedative and hypnotics use, improvement in sleep maintenance, Hamilton Depression Scale (HAMD-17) score, Hamilton Anxiety Scale (HAMA-14) score, Flinders Fatigue Scale (FFS) score, and constitution classification/insomnia pattern score of traditional Chinese medicine, as well as the occurrence of adverse events after 4 weeks' treatment, and follow-up at 8 weeks and 12 weeks.

The main questions it aims to answer are:

1. Are there any significant differences between groups regarding changes in Pittsburgh Sleep Quality Index (PSQI) score, Insomnia Severity Index (ISI) score, subjective sleep latency, sedative and hypnotics usage, improvement in sleep maintenance, Hamilton Depression Scale (HAMD-17) score, Hamilton Anxiety Scale (HAMA-14) score, Flinders Fatigue Scale (FFS) score, and constitution classification/insomnia pattern score of traditional Chinese medicine after 4 weeks' treatment, and follow-up at 8 weeks and 12 weeks.
2. Is the Compound Ciwujia Granules a safe method for chronic insomnia treatment in adults?

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants were adults aged 40-75 years who had insomnia disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition [DSM5]);
2. self-reported history of disturbed sleep (i.e, all the following: ≥30 min to fall asleep, ≥30 min awake during sleep time, and self-reported total sleep time of ≤6·5 h) on at least three nights per week for at least 3 months before screening;(3) diagnosis of "deficiency of the heart and the spleen pattern" or "Qi deficiency of the heart and gallbladder pattern" according to the guidelines for Integrated Traditional Chinese and Western Medicine Treatment of Insomnia Disorders 2023;

(4) baseline Pittsburgh Sleep Quality Index (PSQI) score ≥ 8.

Exclusion Criteria:

1. self-reported allergy symptoms to any of the ingredients;
2. serious physical sickness;
3. a history of suicidal ideation or attempt, acute or chronic psychiatric condition not controlled by therapy;
4. baseline HAMD-17 score ≥17 or HAMA-14 score ≥14;
5. pregnant women;
6. history of drugs or alcohol abuse/dependence;
7. presence of other sleep disorders including sleep apnoea, restless legs syndrome;
8. night, morning or rotating shift work;
9. participation in concurrent clinical trials.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) score | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks and 12 weeks.
  PSQI score, 0-21, and higher scores mean a poorer sleep quality.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) score | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks and 12 weeks.
  ISI score, 0-28, and higher scores mean a worse sleep problem
Hamilton Depression Scale (HAMD-17) score | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks and 12 weeks
  HAMD-17 score, 0-55, and higher scores mean more severe depression.
Hamilton Anxiety Scale (HAMA-14) score | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks and 12 weeks.
  HAMA-14 score, 0-56, and higher scores mean more severe anxiety
Flinders Fatigue Scale (FFS) score | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks and 12 weeks
  FFS score, 0-31, and higher scores mean more severe fatigue
Occurrence of adverse events | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks and 12 weeks.

OTHER OUTCOMES:
Sleep diary | From enrollment to the end of treatment at 4 weeks
  Providing daily information on subjective sleep onset latency, subjective total sleep time, subjective sleep quality, subjective wake after sleep onset, and subjective number of awakenings.
Constitution classification of traditional Chinese medicine | From enrollment to the end of treatment at 4 weeks
  Constitution classification score of traditional Chinese medicine, 0-100, and higher scores mean more likely to have the specified constitution classification.
Insomnia pattern score of traditional Chinese medicine | From enrollment to the end of treatment at 4 weeks
  Insomnia pattern score of traditional Chinese medicine, 0-41, and higher scores mean a worse sleep problem
Use of sedatives and hypnotics | From enrollment to the end of treatment at 4 weeks, and follow-up at 8 weeks, and 12 weeks.
  If it exists, provide information on the use of sedatives or hypnotics (e.g. drug names, dose, and duration)

IPD SHARING:
Plan to Share IPD: No